CLINICAL TRIAL: NCT01648569
Title: Proper Extent of Surgery for Papillary Microcarcinoma
Brief Title: Long-term Outcomes of Total Thyroidectomy Versus Less Than Total Thyroidectomy for Papillary Thyroid Microcarcinoma
Status: Completed | Type: Observational
Sponsor: Korean Association of Endocrine Surgeons (Network)
Responsible Party: Principal Investigator, Jandee Lee, MD PhD, Korean Association of Endocrine Surgeons
Other Study IDs: KoreanAES003
Record Dates: First submitted 2012-07-18; First posted 2012-07-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Papillary Thyroid Microcarcinoma
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Although the vast majority of patients with Papillary Thyroid Microcarcinoma (PTMC) have excellent long-term outcomes, some patients experience tumor recurrence, either locally or, less frequently, as distant metastases, with some patients dying due to this disease. The natural course of PTMC has not always been universally accepted, thus creating controversy concerning the diagnosis and treatment of PTMC. Further, it is not yet possible to confidently identify PTMCs that would take aggressive courses if left untreated. Treatment recommendations range from observation alone to vigorous intervention featuring total thyroidectomy, prophylactic cervical lymph node dissection, and adjuvant RI ablation. Therefore, no consensus has yet been reached on the biological aggressiveness of PTMC or on which therapy is the most appropriate. Moreover, the impact of several clinicopathologic risk factors, including tumor size, is unclear, although patients with tumors ≤ 0.5cm in diameter may have a better prognosis than patients with tumors 0.5-1 cm in size.

Most studies evaluating the proper extent of surgery for PTMC have been retrospective in design. A prospective, long-term, randomized study in a large number of patients, however, may not be feasible owing to the need for an extensive follow-up duration, the costs associated with such a study, and, particularly, its ethical constraints. Consequently, it is not currently possible to determine the prognosis of patients with PTMC or the proper therapeutic approach in these patients. The investigators therefore compared long-term outcomes after total thyroidectomy (TT: total or near-total thyroidectomy) or less than total thyroidectomy (LT: lobectomy or subtotal thyroidectomy) in a large cohort of patients with PTMC, using propensity-score matching to adjust for the uncontrolled assignment of surgical extent in these patients. In addition, the investigators evaluated whether tumor size, ≤ 0.5 cm or > 0.5 cm, had a significant impact in determining the extent of surgery in patients with PTMC.

DETAILED DESCRIPTION:
Study population From March 1986 to December 2006, a total of 5042 patients with PTC (of all tumor sizes) underwent initial surgical therapy at our institution. Of these, 2441 patients (48.4%) had PTMCs ≤ 1 cm in diameter, with 1270 undergoing TT and 1171 undergoing LT. Complete follow-up data for major clinical events were available for 2014 patients (82.5%), including 1015 (79.9%) of the TT group and 999 (85.3%) of the LT group (p=0.083). Patients were followed-up for a median 11.8 years (range, 5 to 26 years). All histopathologic diagnoses were reviewed and verified by endocrine pathologists using WHO criteria. The study protocol was approved by our Institutional Review Board. Details of patients' presentations, surgical and pathologic findings, and adjunctive treatments were obtained from the Yonsei University Thyroid Cancer Database.

Management strategy In patients diagnosed with PTMC after a complete radiologic and histologic examination, the extent of thyroidectomy and radioactive iodine (RI) therapy were based on prognostic factors. However, the protocol of our institution as to how PTMC should be appropriately managed has been changed according to update of clinical reports and validated treatment guidelines. Therefore, the lack of a standardized approach during the study period allowed us to assess the impact of various therapeutic modalities, especially extent of thyroidectomy, in patients with PTMC.

ELIGIBILITY:
Inclusion Criteria:

* From March 1986 to December 2006, a total of 5042 patients with PTC (of all tumor sizes) underwent initial surgical therapy at our institution. Of these, 2441 patients (48.4%) had PTMCs ≤1 cm in diameter, with 1270 undergoing TT and 1171 undergoing LT. Complete follow-up data for major clinical events were available for 2014 patients (82.5%), including 1015 (79.9%) of the TT group and 999 (85.3%) of the LT group (p=0.083). All histopathologic diagnoses were reviewed and verified by endocrine pathologists using WHO criteria.

Exclusion Criteria:

* Patients with follow-up loss

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We evaluated 2014 patients with PTMC who underwent TT (n=1015) or LT (n=999) between March 1986 and December 2006 and for whom complete follow-up data were available for at least 5 years (median 11.8 years; range 5-26 years).
Sampling Method: Non-Probability Sample
Enrollment: 2014 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Overall survival in patients with papillary thyroid microcarcinoma | Overall survival (10-year)
  We analyzed overall survival in patients with PTMC. We also compared the overall survival between total thyroidectomy group versus less than total thyroidectomy group. Survival curves were constructed using the Kaplan-Meier method and compared using the log-rank test.

SECONDARY OUTCOMES:
Disease-free survival in patients with papillary thyroid microcarcinoma | Disease-free survival (10-year)
  We analyzed disease-free survival in patients with PTMC. We also compared the disease-free survival between total thyroidectomy group versus less than total thyroidectomy group. Survival curves were constructed using the Kaplan-Meier method and compared using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Woong Youn Chung, Study Chair — Yonsei University
Locations (1):
- Yonsei University College of Medicidine, Seoul, South Korea